CLINICAL TRIAL: NCT01780610
Title: The Effects of Two Endometrium Preparation Protocols in Frozen-thawed Embryo Transfer in Women With Irregular Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qingxue Zhang, professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SunYatsenU2H- QZhang
Record Dates: First submitted 2013-01-24; First posted 2013-01-31 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Infertility
Keywords: endometrium preparation protocols; frozen-thawed embryo transfer; irregular cycle; randomized controlled trial
MeSH Terms: conditions — Infertility | interventions — Letrozole; Chorionic Gonadotropin; Estradiol; Progesterone; 4-pregnene-3,20-dione

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group OI-A (Other): Patients with irregular cycles undergoing FET in reproductive medicine renter of Sun Yat-sen Memorial Hospital will be recruited , who should not be elder than 40 and had more than 3 frozen embryos.They will be randomized to receive the Letrozole and human chorionic gonadotrophin ovulation induced cycles.
  Interventions: Drug: Letrozole and human chorionic gonadotrophin
- group HRT-B (Other): Patients with irregular cycles undergoing FET in reproductive medicine renter of Sun Yat-sen Memorial Hospital will be recruited, who should not be elder than 40 and had more than 3 frozen embryos will be randomized to receive the estradiol and progesterone replacement therapy cycles.
  Interventions: Drug: estradiol and progesterone

INTERVENTIONS:
Drug: Letrozole and human chorionic gonadotrophin — the follicular development is supported by Letrozole(LE) 2.5mg,once daily is introduced on cycle day 3 .And on cycle day 10 , a Vagina ultrasound is introduced to monitor the development of the follicular ,following by intramuscular gonadotrophin 37.5~75 IU/d until there is a Luteinizing Hormone(LH) surge or ovulation .On the day appearing Luteinizing Hormone surge，patients is always introduced intramuscular human chorionic gonadotrophin(HCG) 10000 IU.If there is sill no Luteinizing Hormone surge when the follicle is 20-24mm ,the ovulation will be induced by HCG.Then the luteum was supported by HCG 2000-2500 IU/3d.Transfer of thawed embryos will be performed 3 days after ovulation is observed.
  Other Names: Letrozole tablets; HCG; Chorionic gonadotrophin; Chorionic gonadotropic hormone
  Arms: group OI-A
Drug: estradiol and progesterone — oral estradiol, 2 mg, once daily, was introduced on cycle day 3 with an increasing doses protocol. If the endometrial thickness was greater than 7mm, progesterone 40-60 mg in oil was administered via intramuscular injection. Transfer of thawed embryos was performed 3 days later
  Other Names: Estradiol Valerate; Progynova; 3,20-pregnene-4; 4-pregnene-3,20-dione; corpus luteum hormone; luteal hormone
  Arms: group HRT-B

SUMMARY:
There are two main cycle regimens used for endometrial preparation for frozen embryo transfer （FET) in women with irregular cycles: hormone replacement therapy cycles (HRT) in which the endometrium is artificially prepared by estrogen and progesterone hormones with/without a gonadotrophin releasing hormone agonist (GnRH-a) down regulation, and ovulation induced cycles (OI) in which follicular development is supported with increasing doses of gonadotrophin hormones and ovulation is induced. At present, there is still no sufficient evidence that which kind of frozen embryo transfer cycle regimen to plan more advantage. The purpose of this study was to compare the pregnancy outcome of hormone replacement therapy cycles (HRT) and ovulation induced cycles (OI) in women with irregular cycles.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial. Patients with irregular cycles undergoing FET in reproductive medicine renter of Sun Yat-sen Memorial Hospital will be recruited who should not be elder than 40 and had more than 3 frozen embryos. They will be randomized to receive either the OI-FET cycle (group OI-A) or the HRT-FET cycle (group HRT-B). In group OI-A, the follicular development is supported by Letrozole(LE) 2.5mg,once daily,is introduced on cycle day 3 .And on cycle day 10 , a Vagina ultrasound is introduced to monitor the development of the follicular ,following by intramuscular gonadotrophin 37.5~75 IU/d until there is a Luteinizing Hormone(LH) surge or ovulation .On the day appearing Luteinizing Hormone surge，patient is always introduced intramuscular human chorionic gonadotrophin(HCG) 10000 IU.If there is sill no Luteinizing Hormone surge when the follicle is 20-24mm ,the ovulation will be induced by HCG.Then the luteum is supported by HCG 2000-2500 IU/3d.Transfer of thawed embryos will be performed 3 days after ovulation is observed. In group HRT-B, oral estradiol, 2 mg, once daily, is introduced on cycle day 3 with an increasing doses protocol. If the endometrial thickness is greater than 7mm, progesterone 40-60 mg in oil will be administered via intramuscular injection. Transfer of thawed embryos will be performed 3 days later.

ELIGIBILITY:
Inclusion Criteria:

* Age forty years old or less
* Has irregular Menstruation (cycle more than 35 days or less than 24 days ) or has regulation Menstruation but previous data suggest that abnormal ovulation
* Frozen embryos number more than three

Exclusion Criteria:

* Has Chocolate cyst or adenomyosis of uterus
* Clear hydrosalpinx
* Uterine scar or intrauterine adhesion and endometrial thickness <7mm before ovulation
* recur thick endometrium（<7mm）
* repeated implantation failure（≥3 times）
* Cancel the cycle because of having no dominant follicle in the ovulation induction（OI)+FET before or the growth of endometrium not good in the HRT+FET before

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 670 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 12 weeks after pregnancy
  12 weeks after pregnancy,people go Vaginal B ultrasonic examination，being saw gestational sac and heart tube beat as ongoing pregnancy

SECONDARY OUTCOMES:
pregnancy rate | 2 weeks after Embryo transplantation
  2 weeks after Embryo transplantation, people go urine HCG and blood HCG test，positive as pregnancy
clinical pregnancy rate | 5 weeks after Embryo transplantation
  5 weeks after Embryo transplantation,people go Vaginal B ultrasonic，being saw the gestation sac as clinical pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Zhang qingxue, doctor, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China